CLINICAL TRIAL: NCT04795427
Title: A Randomized, Open-label, Multi-center, Phase II Study of Asciminib Versus Best Available Therapy in Chinese Patients With Chronic Myelogenous Leukemia in Chronic Phase (CML-CP), Previously Treated With 2 or More Tyrosine Kinase Inhibitors
Brief Title: Study of Efficacy and Safety of CML-CP Patients Treated With Asciminib Versus Best Available Therapy, Previously Treated With 2 or More Tyrosine Kinase Inhibitors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CABL001A2202
Record Dates: First submitted 2021-03-10; First posted 2021-03-12 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Leukemia, Chronic Myelogenous
Keywords: Chronic Myelogenous Leukemia in chronic phase; Chronic Myelogenous Leukemia; CML-CP; Chronic; Chronic Phase; ABL001; asciminib; prior treatment with 2 or more tyrosine kinase inhibitors (TKIs); major molecular response; MMR; Chinese patients; phase ll; open label; best available therapy; BAT
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Bronchiolitis Obliterans Syndrome | interventions — asciminib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- asciminb arm (Experimental): Patients will receive asciminib (40 mg BID continuous)
  Interventions: Drug: asciminib
- best available treatment arm (Experimental): Patients will receive best available therapy chosen by investigator
  Interventions: Other: best available treatment

INTERVENTIONS:
Drug: asciminib — Asciminib comes in 20 mg and 40 mg tablets and is taken orally twice daily
  Other Names: ABL001
  Arms: asciminb arm
Other: best available treatment — Best available treatment will be based on investigator's choice identified prior to randomization. Dose and frequency will depend on label and institutional guidelines for various BAT
  Arms: best available treatment arm

SUMMARY:
The purpose of this Chinese bridging study is to evaluate the efficacy, safety, tolerability and pharmacokinetics of asciminib versus best available therapy in Chinese patients with Chronic Myelogenous Leukemia in chronic phase, previously treated with 2 or more tyrosine kinase inhibitors to support related indication registration in China.

The primary objective of the study is to evaluate the Major Molecular Response (MMR) rate of asciminib treatment at 24 weeks.

DETAILED DESCRIPTION:
The purpose of this Chinese bridging study is to evaluate the efficacy, safety, tolerability and pharmacokinetics (PK) of asciminib versus best available therapy (BAT) in Chinese patients with Chronic Myelogenous Leukemia in chronic phase (CML-CP), previously treated with 2 or more tyrosine kinase inhibitors (TKIs) to support related indication registration in China.

This study will enroll the participants 1) who failed their most recent TKI therapy by meeting the definition of treatment failure as per the 2013 European Leukemia Net (ELN) guidelines, or 2) who were intolerant to the most recent TKI therapy and must have BCR-ABL1 ratio > 0.1% IS at screening.

Eligible participants will be randomized into asciminib arm or the BAT arm on a 2:1 ratio, to receive asciminib treatment (continuous 40 mg BID) or BAT from Day 1 until the end of study treatment period defined as 96 weeks after the last participant receives the first dose.

ELIGIBILITY:
Inclusion Criteria:

Diagnosed as CML-CP:

1. Participants must meet all of the following laboratory values at the screening visit:

   < 15% blasts in peripheral blood and bone marrow < 30% blasts plus promyelocytes in peripheral blood and bone marrow < 20% basophils in the peripheral blood
   * 50 x 10^9/ L (≥ 50,000/mm3) platelets Transient prior therapy related thrombocytopenia (< 50,000/mm3 for ≤ 30 days prior to screening) is acceptable No evidence of extramedullary leukemic involvement, with the exception of hepatosplenomegaly
2. Prior treatment with a minimum of 2 prior ATP-competitive TKIs.
3. Failure (adapted from the 2013 European Leukemia Net (ELN) Guidelines) or intolerance to the most recent TKI therapy at the time of screening.
4. Evidence of typical BCR-ABL1 transcript [e14a2 and/or e13a2] at the time of screening which are amenable to standardized RQ-PCR quantification

Exclusion Criteria:

1. Known presence of the T315I mutation at any time prior to study entry
2. Known second chronic phase of CML after previous progression to AP/BC
3. Previous treatment with a hematopoietic stem cell transplantation
4. Participants planning to undergo allogeneic hematopoietic stem cell transplantation
5. Cardiac or cardiac repolarization abnormality, including any of the following:

   History within 6 months prior to starting study treatment of myocardial infarction, angina pectoris, coronary artery bypass graft Clinically significant cardiac arrhythmias , complete left bundle branch block, high-grade AV block QTcF at screening ≥450 msec (male participants), ≥460 msec (female participants)

   Long QT syndrome, family history of idiopathic sudden death or congenital long QT syndrome, or any of the following:

   Risk factors for Torsades de Pointes including uncorrected hypokalemia or hypomagnesemia, history of cardiac failure, or history of clinically significant/symptomatic bradycardia Concomitant medication(s) with a "Known risk of Torsades de Pointes" that cannot be discontinued or replaced 7 days prior to starting study drug by safe alternative medication.

   Inability to determine the QTcF interval
6. History of acute pancreatitis within 1 year of study entry or past medical history of chronic pancreatitis

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2023-05-29 (Actual); Study Completion 2024-11-18 (Actual)

PRIMARY OUTCOMES:
Major molecular response rate of asciminib | week 24
  Evaluate the major molecular response rate at 24 weeks in asciminib arm

SECONDARY OUTCOMES:
Cytogenetic response (CyR) rate | 24, 48, 96 weeks
  Evaluate the cytogenetic response rate (Complete, Partial, Major, Minor, Minimal, no response) at and by all scheduled data collection time points including 24, 48 and 96 weeks for both asciminib arm and best available treatment arm.
Major molecular response rate of best available treatment arm | week 24
  Evaluate the major molecular response rate at week 24 of best available treatment arm, and compare with asciminib arm
Major molecular response rate of both asciminib arm and BAT armn time points | Up to all participants received at least 96 weeks of randomized study treatment, except week 24
  Evaluate the major molecular response rate, collected at all scheduled data collection time point (except week 24)
major molecular response rate by all scheduled data collection time points | Up to all participants received at least 96 weeks of randomized study treatment
  Evaluate the major molecular rate by all scheduled data collection time points including 24, 48 and 96 weeks by treatment group
Time to major molecular response rate | Up to all participants received at least 96 weeks of randomized study treatment
  Evaluate the time from the date of the first dose of study drug to the date of the first documented MMR by treatment group
Duration of major molecular response | Up to all participants received at least 96 weeks of randomized study treatment
  First document major molecular response to loss of MMR up to 96 weeks after last participant receive the first dose
Overall survival | Up to all participants received at least 96 weeks of randomized study treatment, plus 30 days for safety follow up
  To evaluate the time from the date of randomization to the date of death (including the survival follow-up period)
Progression free survival | Up to all participants received at least 96 weeks of randomized study treatment, plus 30 days for safety follow up
  Evaluate the time from the date of randomization to the earliest occurrence of documented disease progression to AP/BC or the date of death from any cause (including progressions and deaths observed during the survival follow-up period)
Pharmacokinetics (PK) parameter of asciminib: Cmax | Week 2 Day 1 (W2D1)
  Characterize PK of asciminib in the Chinese CML-CP population. Cmax is the maximum (peak) observed plasma drug concentration after dose administration (ng/mL).
PK parameter of asciminib: Tmax | Week 2 Day 1 (W2D1)
  Characterize PK of asciminib in the Chinese CML-CP population. Tmax is the time to reach maximum (peak) plasma drug concentration after dose administration (hr).
PK parameter of asciminib: Ctrough | Week 2 Day 1 (W2D1)
  Characterize PK of asciminib in the Chinese CML-CP population. Trough plasma concentrations (Ctrough)
PK parameter of asciminib: AUCtau | Week 2 Day 1 (W2D1)
  Characterize PK of asciminib in the Chinese CML-CP population. The partial area under the plasma concentration-time curve from dose time to tau (ng*hr/mL). For a bid regimen, Tau=12h.
PK parameter of asciminib: AUClast | Week 2 Day 1 (W2D1)
  Characterize PK of asciminib in the Chinese CML-CP population. AUClast is the The AUC from the time of dosing to the time of the last measurable plasma concentration (Tlast) (ng*hr/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (18):
- China (18):
  - Novartis Investigative Site, Chongqing, Chongqing Municipality
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Shenzhen, Guangdong
  - Novartis Investigative Site, Zhengzhou, Henan
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Nantong, Jiangsu
  - Novartis Investigative Site, Suzhou, Jiangsu
  - Novartis Investigative Site, Nanchang, Jiangxi
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Xian, Shanxi
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Wenzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Shenyang
  - Novartis Investigative Site, Tianjin

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com